CLINICAL TRIAL: NCT07133373
Title: Short Term Turkish Coffee Consumption Elevates Cardiovascular Risk Markers, Decreases Leptin Hormone Levels, and Impairs Sleep Quality in Healthy Young Women: A Pilot Randomized Controlled Trial
Brief Title: Effects Of Turkish Coffee Consumption On Cardiovascular Markers And Sleep In Healthy Women
Acronym: TURCOFFEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Petra (Other)
Responsible Party: Principal Investigator, Nour Amin Elsahoryi, Amman. Jordan, University of Petra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPetra; E/H/5/10/2024 (Other: the Research Ethics Committee of the Faculty of Pharmacy and Medical Sciences at the University of Petra, Amman, Jordan)
Record Dates: First submitted 2025-08-05; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Effects of Turkish Coffee Consumption on Cardiovascular Markers and Sleep in Healthy Women; Cardiometabolic Health Markers, Appetite-regulating Hormones, Inflammation, and Sleep Quality in Healthy Women
Keywords: Turkish coffee; caffeine; young female; cardiovascular health; insomnia; appetite
MeSH Terms: conditions — Inflammation; Sleep Initiation and Maintenance Disorders | interventions — Diagnosis-Related Groups

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel randomized controlled trial. Participants were randomly assigned to either the intervention group (consuming Turkish coffee daily for 4 weeks) or the control group (no coffee consumption). Both groups were followed in parallel during the study period.
Masking Description: No blinding was implemented. Both participants and researchers were aware of group assignment due to the nature of the intervention (coffee consumption).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standardized Turkish coffee (unfiltered and boiled) was administered once daily for 4 weeks. Each serving was approximately 75 mL, prepared using a consistent protocol without added sugar or milk. The coffee was sourced from the same batch and brewed in a traditional cezve. Compliance and adverse effects were monitored throughout the intervention.
  Interventions: Other: Turkish Coffee (unfiltered, boiled)
- control (No Intervention): Participants assigned to the control group were instructed to avoid all forms of coffee for the duration of the 4-week intervention period. They did not receive any dietary or behavioral instructions beyond abstaining from coffee consumption.

INTERVENTIONS:
Other: Turkish Coffee (unfiltered, boiled) — Standardized Turkish coffee (unfiltered and boiled) was administered once daily for 4 weeks. Each serving was approximately 75 mL, prepared using a consistent protocol without added sugar or milk. The coffee was sourced from the same batch and brewed in a traditional cezve. Compliance and adverse effects were monitored throughout the intervention.
  Other Names: case group
  Arms: Intervention

SUMMARY:
This randomized controlled trial aims to evaluate the short-term effects of daily unfiltered Turkish coffee consumption on cardiovascular parameters, appetite-regulating hormones, glucose metabolism, inflammatory markers, and sleep quality in healthy young women. Forty participants will be randomly assigned to an intervention group, consuming standardized servings of Turkish coffee for four weeks, or to a control group abstaining from coffee during the same period. Measurements will be taken at baseline and after the intervention, including blood pressure, lipid profile, leptin, ghrelin, glucose metabolism markers, inflammatory biomarkers, body composition, and sleep quality indices.

DETAILED DESCRIPTION:
Study Design and Participants This study was a pilot randomized, controlled, parallel-group clinical trial to examine the physiological impact of TC consumption over a four-week intervention period among healthy young women. The study was approved by the Institutional Review Board (IRB) at the University of Petra (UOP) with the ID E/H/5/10/2024.

The present study was retrospectively registered at the Open Science Framework (OSF, DOI 10.17605/OSF. IO/2V96N) because OSF is a free and open-access platform that allows transparency and academic cooperation and helps to share the research evaluation process https://osf.io/2v96n/?view_only=19a4815ef45f4ae0814c5a381071163b. This pilot study adhered to the ethical principles of the Declaration of Helsinki following the CONSORT 2010 guidelines for reporting randomized clinical trials, ensuring methodological rigor and transparency, a complementary checklist of CONSORT 2010 is provided supplementary file. After the aims and procedures of the study and the possible risks and rights of the research participants were explained, written informed consent was obtained from all participants. The study duration consisted of conducting participant recruitment and four-week interventions within a two-month period from August 2024 to October 2024.

A total of 50 healthy young females were initially recruited through digital advertisements, social media platforms, and printed flyers. The screening procedures involved a 20-minute face-to-face structured interview to assess eligibility and collect demographic and health-related data. The inclusion criteria were as follows: age (18-25 years), normal body mass index (BMI) (18.5-24.9 kg/m²), nonsmoking status, and infrequent caffeine intake (defined as ≤1 cup/week). Participants with chronic illnesses (e.g., diabetes, thyroid disorders, cardiovascular, or renal conditions), current medication or supplement use affecting appetite, metabolism, or sleep, as well as those following therapeutic diets or enrolled in other clinical trials, were excluded because they met the criteria for prior coffee intervention trials. Those who self-reported as healthy and who met the inclusion were chosen. To control for residual caffeine effects and standardize baseline conditions, a three-week caffeine washout phase was implemented prior to the intervention. During this period, participants were instructed to avoid all caffeine-containing products (coffee, tea, chocolate, soft drinks, energy drinks, and supplements). Adherence was verified through daily self-report logs and unannounced follow-up calls. It is the same strategy, as the previous coffee intervention study protocols washout adherence was used on the basis of subject instruction and self-observation. Three participants (n=3) who consumed caffeine during this phase were excluded from the study.

Following successful washout, 47 participants remained eligible and were randomized via stratified block randomization (based on BMI) into either the intervention group (TC) or the control group. However, prior to initiating the intervention, seven participants (n=7) withdrew voluntarily for personal reasons or scheduling conflicts. The final sample that commenced the intervention comprised 40 participants: 20 assigned to the TC group and 20 assigned to the control group, as shown in Figure 1. The randomization sequence was generated via Randomization.com and administered by an independent researcher to maintain allocation concealment and reduce selection bias.

2.2. Intervention protocol and coffee samples After the washout period and randomization, participants in the intervention group were given a directive to drink TC daily for a period of four weeks, whereas participants in the control group discontinued intake of TC (abstinence) and continued with their usual diet and lifestyle. Owing to the nature of the intervention, blinding was feasible, as it is not possible to find an alternative drink similar in its sensory attributes such as color, smell and flavor that mimics the attributes of the traditional Turkish coffee to use it as a placebo. However, all participants followed the same standardized instructions not to drastically modify dietary patterns during the study. In this study, a sufficient quantity of finely ground Brazilian Arabica TC, consisting of an equal blend of medium and dark roasted coffee beans (5 grams each), was purchased. This is the type of coffee commonly consumed by Jordanian consumers, as reported in studies on Jordanian coffee preparation and drinking habits. The desired amount was distributed to each participant for a period sufficient for the study period, along with optimal storage, preparation, and consumption instructions. The traditional Jordanian way of preparing Turkish coffee was followed by mixing 5 grams of finely ground coffee steeped in 55 mL of cold water in a Rakwa (traditional Turkish coffee pot). The foam on the surface was formed by heating the mixture slowly over low heat. The same amount of boiled plum was approximately 40 mL/serving, as per the national standard consumption size. The caffeine content and bioactive compound exposure per cup were calculated using this standardized serving volume. To approximate daily consumption habits and maintain the integrity of coffee components, this unfiltered preparation method was used while preserving bioactive compounds, such as chlorogenic acids and diterpenes. Each participant consumed three daily cups (40 mL each) of TC throughout the day over three specified time periods: the first cup between 7 and 9 AM, the second cup between 12 and 2 PM, and the third cup between 3 and 4 PM, with evening consumption strictly prohibited. The study adopted this protocol through morning, midday and early-afternoon coffee consumption because research has shown that caffeine consumed 6 h before bedtime disrupts sleep quality. Infinitely tracked protocol compliance through daily logs and calls to its participants. The beverage was consumed with no additives (except where the subjects habitually used sugar, these subjects continued their habitual sugar quantity to avoid changing their habitual consumption). Coffee packets were preportioned, and each participant was given preparation instructions along with calibrated utensils to ensure standardization and compliance. In the laboratory, the caffeine concentration in the prepared coffee solution was analyzed and determined to be approximately 1.77 mg/mL via high-performance liquid chromatography (HPLC) coupled with a diode array detector (DAD) and mass spectrometer (MS) and was found to be equivalent to approximately 71 mg of caffeine/40 mL cup. This approach was consistent across all consumed servings and permitted precise quantification of the bioactive load. Daily intake logs and random follow-up phone calls were used to monitor participant compliance. Furthermore, at baseline and postintervention, 24-hour dietary recall was standardized through statistical analysis for potential confounding variables such as physical activity and dietary intake.

2.3. Blood collection and biomarker assessment Blood samples were collected at baseline (week 0) and after the fourth week of intervention (week 4) of the study, during a fasting period of at least 10 h after overnight fasting. A certified phlebotomist drew venous blood from the antecubital vein via sterile and standardized protocols. All samples were centrifuged at 4°C and 3000 rpm for 10 min immediately following collection to separate the serum and plasma. First, aliquots were stored at -80°C until further laboratory analysis.

2.4. Metabolic and glycemic biomarkers Fasting blood glucose (FBS) was measured via the TRUE METRIX® Meter Starter Kit, which employs electrochemical biosensor technology and provides fast, point-of-care results with a four-second reading time and minimal sample volume (0.5 µL). Glycated hemoglobin (HbA1c), representing longer-term glycemic control, was assessed via the HP-AFS/1-PLUS analyzer (Hitachi), which integrates nephelometry, turbidimetry, and immunofluorescence technologies for increased measurement sensitivity.

2.5. Lipid Profile and Cardiovascular Risk Indicators The same HP-AFS/1-PLUS system was used to analyze the lipid biomarkers total cholesterol, triglyceride (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C). Resting SBP, DBP and HR were measured at both time points via a validated and calibrated Omron M7 Intelli IT (HEM-7361T-EBK) automatic sphygmomanometer to determine cardiovascular effects. All the measurements were carried out in a clinical environment after the subjects had been seated for at least five minutes and had rested. The right arm was read in triplicate and averaged to ensure reliability and reduce variability.

2.6. Assessment of Appetite Biomarkers Serum leptin and ghrelin levels were measured before and after the intervention to study appetite regulatory mechanisms. The quantification of these hormones was carried out with validated nephelometric and immunofluorescence-based protocols via an HP-AFS/1-PLUS analyzer. The role of leptin as a satiety signal and ghrelin as a hunger signal, when combined, helps gain some insight into how people react in regard to energy regulation and how coffee intake is one aspect that plays a part in this process.

2.7. Assessment of Inflammation Biomarkers The biomarkers of inflammation (C-reactive protein (CRP) and tumor necrosis factor-alpha (TNF-α)) were measured at baseline and after intervention. Blood samples taken the next morning, following an overnight fast, were centrifuged to separate the serum. The levels of CRP in high-sensitivity immunoturbidimetric assay (mg/L), whereas the levels of TNF-alpha of high-sensitivity enzyme-linked immunosorbent assay (ELISA) kit with a detection range of 15.631000 pg/mL. The readings of absorbances were taken using a BioTek Epoch™ 2 Microplate Spectrophotometer (Agilent Technologies, USA) with Gen 5™ software to analyze and retrieve the data. All of them were performed according to the instructions of the manufacturers. The validated analysis methods employed are reported in similar intervention trial [31].

2.8. Dietary Intake A single 24-h dietary recall was used to assess dietary intake during the intervention period. This strategy was selected as feasible and to ease participant burden while habitual intake was surveyed. A trained researcher conducted the recall interview and recorded all the food and beverage items they consumed in the past 24 hours, including portion size, preparation method and time of consumption. The macronutrients and micronutrients were estimated accurately via the ESHA Food Processor (version 8.6), which was used to analyze the data. A single 24-h recall has limitations in assessing habitual diet; however, it provides a suitable method to control potential acute dietary confounders across study groups in this short-term intervention.

2.9. Insomnia assessment The Arabic version of the Insomnia Severity Index (ISI) was utilized to assess insomnia symptoms at baseline and after the intervention. ISI used in this study was already being translated and validated as Insomnia Severity Index in Arabic population. It was shown to be of acceptable internal consistency (Cronbach alpha 0.84) and high convergent validity with PSQI (zero order correlation coefficient r = 0.76, p < 0.001). The Sleep Difficulties and Daytime Functioning Severity Scale is a 7-item, self-administered measure that assesses the severity of sleep difficulties as well as the impact of sleep difficulties on daytime functioning. The Arabic version of the ISI has been culturally adapted and validated for use among Arabic-speaking populations with respect to linguistic and psychometric consistency. A total score between 0 and 28 is obtained by giving each item a score of 0 to 4 (no problem) to 4 (very severe). Insomnia severity was defined as ranging from 0-7 (no insomnia), 8-14 (subthreshold), 15-21 (moderate), or 22-28 (severe). The measurement was performed at both time points via the same standardized tool to ensure consistent measurement.

2.10. Body composition assessment A set of initial screening visit measures were collected for baseline anthropometric parameters as part of determining eligibility on the basis of body composition. Whole-body and segmental components such as fat mass, fat-free mass, total body water, and skeletal muscle mass were estimated via the InBody 970 Body Composition Analyzer (Model 1421000139, InBody Co., Ltd., Seoul, Republic of Korea) via multifrequency bioelectrical impedance analysis (BIA). The measurement accuracy and reproducibility were achieved by regularly calibrating the device in accordance with the manufacturer's specifications. Assessments were performed in the early morning, after a minimum of 10 h of overnight fasting and prior to any study-related interventions to reduce the potential of variability resulting from the last food intake. They were provided instructions to prevent alcohol and strenuous physical activity for 24 h prior and to stay well hydrated but not to overload fluids. All metallic items were removed, and clothing was standardized prior to measurement. Where not possible, measurements were scheduled during the follicular phase of the menstrual cycle, as this aligns with best practices of BIA research in female participants in an effort to minimize hormonal effects on fluid distribution and body composition. The body composition data collected were used as the baseline reference and for tracking any physiological changes during and after the four weeks of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Healthy female participants aged between 18 and 35 years

Body Mass Index (BMI) between 18.5 and 29.9 kg/m²

Habitual coffee consumers (1-2 cups/day)

Not on a weight-loss or special medical diet

Not taking medications or supplements that affect sleep, appetite, metabolism, or cardiovascular function

Non-smokers and not using recreational drugs

Willing to comply with study protocol and attend all assessments

Exclusion Criteria:

Pregnancy or lactation

Diagnosed chronic diseases (e.g., diabetes, hypertension, cardiovascular disease)

Known sleep disorders or psychological conditions

Allergy or sensitivity to coffee or caffeine

Irregular menstrual cycle or hormonal disorders

Shift workers or frequent travelers across time zones

Participation in other clinical trials within the past 3 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure after 4 weeks of Turkish coffee consumption | Baseline and Week 4
  Systolic and diastolic blood pressure were measured at baseline and after 4 weeks using a validated electronic monitor (Omron M6). Participants were seated in a relaxed position, and the average of two readings was recorded. The change in blood pressure levels was used to assess cardiovascular effects of Turkish coffee consumption.

SECONDARY OUTCOMES:
Change in serum leptin and ghrelin levels after 4 week | Baseline and Week 4
  Blood samples were collected at baseline and at the end of the intervention to assess serum leptin and ghrelin concentrations using ELISA kits.

CONTACTS AND LOCATIONS:
Locations (1):
- UOP, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared due to confidentiality concerns and ethical limitations related to the nature of the data collected. The data include sensitive health and behavioral variables that cannot be adequately de-identified.